CLINICAL TRIAL: NCT04781881
Title: Special Drug Use Surveillance for Entresto Tablets (Chronic Heart Failure, CLCZ696B1401)
Brief Title: Special Drug Use Surveillance for Entresto Tablets
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696B1401
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; Entresto; Japan; sacubitril/valsartan; sacubitril valsartan sodium hydrate
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Entresto: Patients administered Entresto by prescription
  Interventions: Drug: Entresto

INTERVENTIONS:
Drug: Entresto — There is no treatment allocation. Patients administered Entresto by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a single arm, multicenter, observational study in Japanese chronic heart failure patients.

DETAILED DESCRIPTION:
This study is a special drug use surveillance to evaluate the safety and efficacy of Entresto Tablets (hereafter called Entresto) clinically administered in Japanese patients for the newly approved indication of "chronic heart failure" and to be conducted as one of the RMP-specified additional pharmacovigilance activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written consent to cooperate in this study before the start of Entresto
* Patients using Entresto for the first time for the following indication Indication: chronic heart failure patients on standard of care for chronic heart failure

Exclusion Criteria:

* Patients with a history of treatment with a drug containing the same ingredient (investigational drug or post-marketing clinical study drug) as Entresto
* The following patients for whom Entresto is contraindicated in the package insert Patients with a history of hypersensitivity to any of the Entresto ingredients Patients with a history of angioedema (angiotensin II receptor blockers or angiotensin converting enzyme inhibitors-induced angioedema, hereditary angioedema, acquired angioedema, idiopathic angioedema etc.) Diabetic patients on aliskiren fumarate Patients with severe hepatic impairment (Child-Pugh class C) Pregnant or possibly pregnant women

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients using Entresto for the newly approved indication of "chronic heart failure"
Sampling Method: Non-Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of Entresto in chronic heart failure patients | Up to 52 weeks
  EAIR of hypotension, hyperkalemia, renal impairment and dehydration will be collected.
  EAIR: n/T, n: total number of events included in the analysis, T(100 patient years): total up-to-event/censoring duration-time summarized over patients

SECONDARY OUTCOMES:
To evaluate the impact of risk factors | Up to 52 weeks
  Subgroup analysis of EAIR (patients/100 patient-years) of hypotension, hyperkalemia, renal impairment and dehydration by risk factor will be presented EAIR: n/T, n: total number of events included in the analysis, T(100 patient years): total up-to-event/censoring duration-time summarized over patients
To investigate the occurrence of AEs, SAEs, ADRs and serious ADRs | Up to 52 weeks
  A SAE is defined as an AE whose description suggests that it is serious or whose outcome is fatal.
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Entresto or whose causality is not recorded
EAIR for each of the clinical events | Up to 52 weeks
  EAIR: n/T, n: total number of events included in the analysis, T(100 patient years): total up-to-event/censoring duration-time summarized over patients
Kaplan-Meier curve for each of the clinical events | Up to 52 weeks
  Kaplan-Meier estimate of cumulative failure rate(%) will be collected
Total frequency of hospitalization due to heart failure | Up to 52 weeks
  Total frequency of hospitalization due to heart failure will be collected
To investigate data on the administration of Entresto in clinical use | Up to 52 weeks
  Data on Entresto administration will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (93):
- Japan (93):
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Nishio, Aichi-ken
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Yatomi, Aichi-ken
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sakura, Chiba
  - Novartis Investigative Site, Yachiyo, Chiba
  - Novartis Investigative Site, Imabari, Ehime
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Kasuya-gun, Fukuoka
  - Novartis Investigative Site, Ukiha, Fukuoka
  - Novartis Investigative Site, Iwaki, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Takasaki, Gunma
  - Novartis Investigative Site, Fuchū, Hiroshima
  - Novartis Investigative Site, Mihara, Hiroshima
  - Novartis Investigative Site, Takehara, Hiroshima
  - Novartis Investigative Site, Abashiri, Hokkaido
  - Novartis Investigative Site, Fukagawa, Hokkaido
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Ishikari, Hokkaido
  - Novartis Investigative Site, Iwamizawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Awaji, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kakogawa, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Mukou-City, Kyoto
  - Novartis Investigative Site, Iga, Mie-ken
  - Novartis Investigative Site, Tamaru, Mie-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Higashimatsushima, Miyagi
  - Novartis Investigative Site, Shiogama, Miyagi
  - Novartis Investigative Site, Saito, Miyazaki
  - Novartis Investigative Site, Iki, Nagasaki
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kita-Katsuragi-gun, Nara
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Urasoe, Okinawa
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Kishima-gun, Saga-ken
  - Novartis Investigative Site, Ureshino, Saga-ken
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Toda, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Higashiohmi, Shiga
  - Novartis Investigative Site, Gotemba, Shizuoka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Nasushiobara, Tochigi
  - Novartis Investigative Site, Utsunomiya, Tochigi
  - Novartis Investigative Site, Adachi City, Tokyo
  - Novartis Investigative Site, Akiruno, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Minato, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nakano City, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Toshima City, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
  - Novartis Investigative Site, Sakata, Yamagata
  - Novartis Investigative Site, Shinjō, Yamagata
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōita
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokushima
  - Novartis Investigative Site, Toyama
  - Novartis Investigative Site, Wakayama
  - Novartis Investigative Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: No